CLINICAL TRIAL: NCT04690283
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase Ⅲ Clinical Trial of Yiqi Wenjing Prescriptions for Preventing Oxaliplatin-induced Peripheral Neuropathy
Brief Title: Yiqi Wenjing Prescriptions Preventive Efficacy of Oxaliplatin-induced Peripheral Neuropathy Clinical Trial
Acronym: YWPPEOPNCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing NingQi Medicine Science and Technology Co., Ltd. (Industry)
Collaborators: Jiangsu Provincial Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Jiangsu Cancer Institute & Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SBE2019750381
Record Dates: First submitted 2020-12-13; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Colorectal Cancer
Keywords: clinical trial; Yiqi Wenjing prescriptions; oxaliplatin-induced peripheral neuropathy; randomized; placebo-controlled
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Subject diagnosed with colorectal cancer stages IIa-IIIc, suitable for receiving FOLFOX4 or mFOLFOX6 as adjuvant chemotherapy after radical resection of colorectal cancer, receiving each dose and cumulative dose of oxaliplatin are 85mg/m2 and ≥540 mg/m2 respectively, with Karnofsky performance status scale (Schag et al.1984) index ≥60 points and an expected survival time ≥6 months, over 18 years of age, men or women, without severe damage of the heart, liver, kidney or hematopoietic system.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo-control group (Placebo Comparator): Subjects will receive FOLFOX4 or mFOLFOX6 or XELOX chemotherapy regimen and placebo treatment twice a day (1/2 bag, morning and evening) for at least three months and one year follow up.
  Interventions: Drug: Mimetic granules of Yiqi-Wenjing prescriptions
- Treatment group I (Experimental): Subjects will receive FOLFOX4 or mFOLFOX6 or XELOX chemotherapy regimen and orally take Huangqi Guizhi Wuwu granules twice a day (1/2 bag, morning and evening) for at least three months and one year follow up.
  Interventions: Drug: Huangqi-Guizhi-Wuwu granules
- Treatment group II (Experimental): Subjects will receive FOLFOX4 or mFOLFOX6 or XELOX chemotherapy regimen and orally take Danggui Sini granules twice a day (1/2 bag, morning and evening) for at least three months and one year follow up.
  Interventions: Drug: Danggui-Sini granules

INTERVENTIONS:
Drug: Mimetic granules of Yiqi-Wenjing prescriptions — The intervention relates to a multiple granules, which contains 2.5% concentrated Huangqi-Guizhi-Wuwu decoction (a classical traditional Chinese prescription consists of astragalus membranaceus, cassia twig, radix paeoniae alba, ginger and jujube), 2.5% concentrated Danggui-Sini decoction (a classical traditional Chinese prescription consists of angelica sinensis, cassia twig, radix paeoniae alba, asarum, tetrapanax papyriferus, jujube and honey-fried licorice root), bitter principle, food colouring and starch.
  Other Names: Mimetic granules of Huangqi-Guizhi-Wuwu plus Danggui-Sini decoction
  Arms: Placebo-control group
Drug: Huangqi-Guizhi-Wuwu granules — The intervention relates to a traditional Chinese prescription granules, which contains astragalus membranaceus, cassia twig, radix paeoniae alba, ginger and jujube.
  Arms: Treatment group I
Drug: Danggui-Sini granules — The intervention relates to a traditional Chinese prescription granules, which contains angelica sinensis, cassia twig, radix paeoniae alba, asarum, tetrapanax papyriferus, jujube and honey-fried licorice root.
  Arms: Treatment group II

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, multicenter phase III clinical trial of Yiqi Wenjing prescriptions for Preventing Oxaliplatin-induced Peripheral Neuropathy.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blind, and multicenter clinical trial. Three hundred sixty postoperative patients with colon cancer stage IIa-IIIc will be randomly assigned into treatment group I, treatment group II and placebo-control group, taking Huangqi Guizhi Wuwu granules, Danggui Sini granules and the mimetic granules of Yiqi Wenjing granules respectively. All subjects will receive mFOLFOX6 or FOLFOX4 or XELOX chemotherapy regimen along with traditional Chinese medicine(TCM) or placebo treatment per day for at least three months and one year follow up. EORTC QLQ-CIPN20 will be used to assess the degree of peripheral neuropathy as the primary outcome measure. Grades of OIPN evaluated by NCI-CTCAE 5.0, quality of life evaluated by EORTC QLQ-C30, chemotherapeutic efficacy evaluated by RESIST 1.1, and the number of completed chemotherapy cycles are selected as the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with colorectal cancer stages IIa-IIIc, confirmed by histopathological examination, according to CSCO guidelines for diagnosis and treatment of colorectal cancer.
* Subject suitable for receiving FOLFOX4 or mFOLFOX6 as adjuvant chemotherapy after radical resection of colorectal cancer, receiving each dose and cumulative dose of oxaliplatin are 85mg/m2 and ≥540 mg/m2 respectively.
* Subject with Karnofsky performance status scale (Schag et al.1984) index ≥60 points and an expected survival time ≥6 months.
* Subject over 18 years of age, men or women.
* Subject without severe damage of the heart, liver, kidney or hematopoietic system.

Exclusion Criteria:

* Subject with any grade of peripheral neuropathy.
* Subject who has ever received treatment of neurotoxic chemotherapeutics, such as oxaliplatin, cisplatin, taxanes, or vinca alkaloids.
* Subject who is receiving agents with potential preventive or therapeutic effects to neuropathy, such as duloxedine, carbamazepine, venlafaxine, gabapentin, pregabalin, phenytoin, valproate, milnacipran, or tricyclic antidepressant.
* Subject who is participating or have participated in other clinical trials.
* Subject with a family history of hereditary/familial neuropathy.
* Subject who cannot take drugs orally.
* Subject with mental illness who cannot cooperate.
* Pregnant or lactation period women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The dynamic change of the degree of oxaliplatin-induced peripheral neuropathy | On 1 day before and 3 days after the beginning of each cycle(each FOLFOX4 or mFOLFOX6 cycle is 14 days, each XELOX cycle is 21 days) up to Cycle 6, 1 month after the end of Cycle 6, and then every 3 months up to 1 year.
  The degree of oxaliplatin-induced peripheral neuropathy will be evaluated according to the score of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty item scale(EORTC QLQ-CIPN20, 20-80 scores, higher scores mean a worse outcome), which is graded by the subject. In order to observe the dynamic change of OIPN, this trial sets multiple measure time points.

SECONDARY OUTCOMES:
The dynamic change of the grades of oxaliplatin-induced peripheral neuropathy | On 1 day before the beginning of each cycle(each FOLFOX4 or mFOLFOX6 cycle is 14 days, each XELOX cycle is 21 days) up to Cycle 6.
  The grades of oxaliplatin-induced peripheral neuropathy will be evaluated according to the grades of National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE 5.0, 0-5 grades, higher grade means a worse outcome), which is graded by the doctor. In order to observe the dynamic change of OIPN, this trial sets multiple measure time points.
The dynamic change of quality of life | On 1 day before the beginning of each cycle(each FOLFOX4 or mFOLFOX6 cycle is 14 days, each XELOX cycle is 21 days) up to Cycle 6.
  Quality of life will be evaluated according to the score of European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30, 28-112 scores, higher scores mean a worse outcome). In order to observe the dynamic change of QOL, this trial sets multiple measure time points.
The number of completed chemotherapy cycles | At the end of Cycle 6 or after the last chemotherapy(each FOLFOX4 or mFOLFOX6 cycle is 14 days, each XELOX cycle is 21 days).
  The number of completed chemotherapy cycles will be recorded. If the result is less then 6, the specific reason should be noted.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for reference include the vague name, gender, age, diagnosis, the type and number of chemotherapy regimens, the degree and grades of oxaliplatin-induced peripheral neuropathy
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting in January 2025 and forever

REFERENCES:
- [Derived] Gu Z, Wei G, Zhu L, Zhu L, Hu J, Li Q, Cai G, Lu H, Liu M, Chen C, Ji Y, Li G, Huo J. Preventive Efficacy and Safety of Yiqi-Wenjing-Fang Granules on Oxaliplatin-Induced Peripheral Neuropathy: A Protocol for a Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial. Evid Based Complement Alternat Med. 2021 Sep 29;2021:5551568. doi: 10.1155/2021/5551568. eCollection 2021. PMID 34630609